CLINICAL TRIAL: NCT03148015
Title: Novel Molecular Targets for Ductal Carcinoma In Situ (DCIS)
Status: Completed | Type: Observational
Sponsor: Sentara Norfolk General Hospital (Other)
Collaborators: George Mason University (Other); Dorothy G. Hoefer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 16-03-EX-0064
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsy or surgical tissue specimen slides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADH/LCIS: Atypical Ductal Hyperplasia or Lobular carcinoma in situ with DCIS
  Interventions: Other: Biomarkers
- DCIS: Pure Ductal Carcinoma in Situ
  Interventions: Other: Biomarkers
- Invasive: invasive ductal carcinoma with DCIS
  Interventions: Other: Biomarkers

INTERVENTIONS:
Other: Biomarkers — Evaluate the intracellular and intraluminal distribution of autophagy and calcium efflux markers in each breast lesion in comparison to the HER2, proliferation (Ki-67, PCNA), p53, inflammatory, and apoptotic (Annexin-1) markers in the same patient. Determine the qualitative amount and localization of PMCA2 and Vitamin D Receptor in each breast lesion with intraductal calcium spicules compared to lesions without microcalcifications.

SUMMARY:
This project is an immunohistochemical study of archived patient breast tissue, specifically pre-invasive lesion specimens. The purpose is the discovery of novel molecular markers of pre-invasive breast lesions. These novel markers, once validated in this study, can serve as targets for individualized prevention therapy, neoadjuvant therapy for ductal carcinoma in situ (DCIS), or predictors of lesion aggressiveness. We have discovered two novel classes of DCIS molecular pathways required for the survival of DCIS neoplastic cells that will serve as the basis for the candidate molecules to be evaluated in this proposed study. The first class of DCIS molecular markers is autophagy, a cell survival mechanism that we discovered to be highly augmented in the hypoxic and nutrient deprived intraductal neoplastic cells of human DCIS (1-4). The second class of biomarker is calcium efflux that is mediated in breast cells by the calcium export pump Plasma Membrane Calcium ATPase (PMCA2) (5, 6). During normal lactation, breast epithelium pumps large concentrations of calcium into milk. In neoplastic lesions, calcium is exported by PMCA2 as a cell survival mechanism, since cells under metabolic stress accumulate calcium to a toxic level. Calcium export in DCIS may also contribute to intraductal calcifications, a hallmark of high grade DCIS and the most common marker of DCIS on mammography (7).

Sentara cares for hundreds of patients per year who are diagnosed with breast pre-invasive lesions, including atypical ductal hyperplasia (ADH), ductal carcinoma in situ (DCIS), and lobular carcinoma in situ (LCIS). Sentara treats 25% of the women with breast cancer in Virginia. Coupled with information from the Sentara Cancer Registry, Dr. Hoefer or a research team member will identify eligible patients with ADH, DCIS, and/or LCIS at the time of the core biopsy diagnosis, surgical therapy, and/or upon lesion recurrence. After receiving written informed consent from the eligible patients, Sentara Pathology will retrieve the corresponding tissue blocks. The recut tissue sections will be processed at George Mason University, Center for Applied Proteomics and Molecular Medicine for markers relevant to calcium signaling, Vitamin D response, proliferation, autophagy and inflammation. Combined with the translational research expertise/technology in the Center for Applied Proteomics and Molecular Medicine at George Mason University, Sentara's diverse patient cohort provides an opportunity to address the most fundamental unanswered questions surrounding the etiology, progression, and therapy of pre-invasive breast lesions.

DETAILED DESCRIPTION:
Sentara Healthcare is a progressive and integrated healthcare organization that cares for hundreds of patients per year who are diagnosed with breast cancer and pre-invasive lesions, including atypical ductal hyperplasia (ADH), ductal carcinoma in situ (DCIS), and lobular carcinoma in situ (LCIS). Sentara Healthcare maintains a Cancer Registry which includes complete clinical information and disposition information of tissue blocks collected at the time of the core biopsy diagnosis, the surgical therapy, and upon lesion recurrence. Combined with the translational research expertise/technology in the Center for Applied Proteomics and Molecular Medicine (CAPMM) at George Mason University (GMU), the Sentara Healthcare extensive patient cohort provides an opportunity to address the most fundamental unanswered questions surrounding over-treatment and under-treatment of pre-invasive breast lesions:

1. Does the histopathologic/molecular character of the carcinoma in situ, the immune infiltrate, and/or the stroma, correlate with the type of lesion (ADH, DCIS or LCIS), the grade of the lesion, or the presence of later recurrence?
2. Does the level of autophagy within the lesion duct, or the level of PMCA2, of the pre-invasive lesion, correlate with lesion grade, the level of apoptosis, or the presence of later recurrence?
3. Does the level of Vitamin D receptor correlate with the level of PMCA2?

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female, at least 18 years of age.
* Patients or their legally authorized representative must have signed and dated an informed consent form
* Patients must have at minimum, adequate samples of breast tissue available for use in this study.
* Patients with a tissue diagnosis of low, intermediate or high grade ductal carcinoma in situ or ductal carcinoma in situ with microinvasion.
* Patients with a diagnosis of atypical ductal hyperplasia, lobular cancer in situ or any preinvasive breast lesion.
* Patients with ductal carcinoma in situ undergoing either lumpectomy and radiation or mastectomy.
* Patients with a diagnosis of invasive ductal cancer.

Exclusion Criteria:

* Male.
* Patients under the age of 18 or over the age of 89.
* Patient desires not to participate in the study.
* Inability to consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18 or older who have had a breast biopsy and or surgery with breast tissue available. Patient must be diagnosed with ADH, DCIS, LCIS or invasive ductal cancer.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Molecular and Histopathologic Characteristics | Duration of Study, estimated 2 years
  Demonstrate the concomitant activation of autophagy and calcium efflux in pre-invasive breast lesions. Compare the molecular and histopathologic characteristics of the breast DCIS/invasive lesion to the lesion microenvironment.

SECONDARY OUTCOMES:
Biomarkers | Duration of Study, estimated 2 years
  Identify and characterize biomarkers in the DCIS breast lesion and invasive that correlate with autophagy, calcium signaling and inflammation.
Histopathologic/Molecular Characteristics by lesion type | Duration of Study, estimated 2 years
  Establish the histopathologic/molecular character of the stroma, the pre-invasive lesion, and correlate with the type of lesion (ADH, DCIS or LCIS), the grade of the lesion, or the presence of invasive carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Sentara Surgery Specialists and Dorothy G Hoefer Comprehensive Breast Center, Newport News, Virginia, United States

IPD SHARING:
Plan to Share IPD: No